CLINICAL TRIAL: NCT04390399
Title: Open-label, Randomized, Comparative Phase 2 Study of Combination Immunotherapy Plus Standard-of-care Chemotherapy Versus Standard-of-care Chemotherapy for the Treatment of Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Combination Immunotherapy Plus Standard-of-Care Chemotherapy Versus Standard-of-Care Chemotherapy for the Treatment of Locally Advanced or Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-88
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ALT-803; 130-nm albumin-bound paclitaxel; Gemcitabine; Cyclophosphamide; Fluorouracil; Leucovorin; irinotecan sucrosofate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A Control Treatment Arm (Active Comparator): SBRT + gemcitabine + nab-paclitaxel
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Procedure: SBRT
- Cohort A Experimental Treatment Arm 1 (Experimental): SBRT + cyclophosphamide + gemcitabine + nab-paclitaxel + aldoxorubicin HCl + N-803
  Interventions: Biological: N-803; Drug: Aldoxorubicin HCl; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Cyclophosphamide; Procedure: SBRT
- Cohort A Experimental Treatment Arm 2 (Experimental): SBRT + cyclophosphamide + gemcitabine + nab-paclitaxel+ aldoxorubicin HCl + N-803 + PD-L1 t-haNK
  Interventions: Biological: N-803; Drug: Aldoxorubicin HCl; Biological: PD-L1 t-haNK; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Cyclophosphamide; Procedure: SBRT
- Cohort B Control Treatment Arm (Active Comparator): Irinotecan liposome + 5-FU/leucovorin
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Irinotecan liposome
- Cohort B Experimental Treatment Arm (Experimental): SBRT + cyclophosphamide + gemcitabine + nab-paclitaxel+ aldoxorubicin HCl + N-803 + PD-L1 t-haNK
  Interventions: Biological: N-803; Drug: Aldoxorubicin HCl; Biological: PD-L1 t-haNK; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Cyclophosphamide; Procedure: SBRT
- Cohort C Experimental Treatment Arm (Experimental): SBRT + cyclophosphamide + gemcitabine + nab-paclitaxel + aldoxorubicin + N-803 + PD-L1 t-haNK
  Interventions: Biological: N-803; Drug: Aldoxorubicin HCl; Biological: PD-L1 t-haNK; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Cyclophosphamide; Procedure: SBRT

INTERVENTIONS:
Biological: N-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
  Arms: Cohort A Experimental Treatment Arm 1; Cohort A Experimental Treatment Arm 2; Cohort B Experimental Treatment Arm; Cohort C Experimental Treatment Arm
Drug: Aldoxorubicin HCl — Aldoxorubicin hydrochloride
  Arms: Cohort A Experimental Treatment Arm 1; Cohort A Experimental Treatment Arm 2; Cohort B Experimental Treatment Arm; Cohort C Experimental Treatment Arm
Biological: PD-L1 t-haNK — PD-L1 t-haNK suspension for infusion
  Arms: Cohort A Experimental Treatment Arm 2; Cohort B Experimental Treatment Arm; Cohort C Experimental Treatment Arm
Drug: Nab-paclitaxel — Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
  Arms: Cohort A Control Treatment Arm; Cohort A Experimental Treatment Arm 1; Cohort A Experimental Treatment Arm 2; Cohort B Experimental Treatment Arm; Cohort C Experimental Treatment Arm
Drug: Gemcitabine — 2', 2'-difluoro 2'deoxycytidine, dFdC
  Arms: Cohort A Control Treatment Arm; Cohort A Experimental Treatment Arm 1; Cohort A Experimental Treatment Arm 2; Cohort B Experimental Treatment Arm; Cohort C Experimental Treatment Arm
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
  Arms: Cohort A Experimental Treatment Arm 1; Cohort A Experimental Treatment Arm 2; Cohort B Experimental Treatment Arm; Cohort C Experimental Treatment Arm
Drug: 5-Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
  Arms: Cohort B Control Treatment Arm
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
  Arms: Cohort B Control Treatment Arm
Procedure: SBRT — Stereotactic Body Radiation Therapy
  Arms: Cohort A Control Treatment Arm; Cohort A Experimental Treatment Arm 1; Cohort A Experimental Treatment Arm 2; Cohort B Experimental Treatment Arm; Cohort C Experimental Treatment Arm
Drug: Irinotecan liposome — Irinotecan hydrochloride trihydrate is (S)-4,11-diethyl-3,4,12,14-tetrahydro-4-hydroxy-3,14-dioxo1H-pyrano[3',4':6,7]-indolizino[1,2-b]quinolin-9-yl-[1,4'bipiperidine]-1'-carboxylate, monohydrochloride, trihydrate
  Arms: Cohort B Control Treatment Arm

SUMMARY:
This is a phase 2, three-cohort (2 randomized and 1 single-arm), open-label study to evaluate the comparative efficacy and overall safety of standard-of-care chemotherapy versus standard-of-care chemotherapy in combination with aldoxorubicin HCl, N-803, and PD-L1 t-haNK in subjects with locally advanced or metastatic pancreatic cancer. Each treatment setting (ie, first line maintenance, second line, or third line or greater) will be evaluated independently as a separate cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Have histologically confirmed unresectable, locally advanced or metastatic pancreatic cancer.

   1. For Cohort A, subjects must have initially received, or are currently receiving, continuous treatment with gemcitabine plus nab-paclitaxel for at least 16 weeks and have confirmed PR, CR, or SD prior to receiving first-line maintenance therapy on this study. Duration of actual initial treatment may be unlimited as long as no evidence of disease progression is noted by the Investigator at the time of randomization.
   2. For Cohort B, subjects must have PD after receiving initial treatment with FOLFOX, FOLFIRINOX, or a gemcitabine- or paclitaxel-based therapy for pancreatic cancer.

      Subjects who discontinued prior therapy due to toxicity, intolerance, or available therapy was clinically contraindicated are allowed.
   3. For Cohort C, subjects must have PD after receiving at least 2 lines of therapy for pancreatic cancer, including but not limited to neoadjuvant, adjuvant, and/or metastatic settings.
4. ECOG PS of 0 or 1.
5. Have at least 1 measurable lesion and/or non-measurable disease evaluable in accordance with RECIST V1.1.
6. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
7. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception while on study and for at least 5 months after the last dose of study treatment. Non-sterile male subjects must agree to use a condom while on study and for up to 5 months after the last dose of study treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, IUDs, oral contraceptives, and abstinence.

Exclusion Criteria

1. Body weight ≤ 40 kg at screening.
2. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
3. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
4. For Cohort A only: tumors harboring germline BRCA1/2 mutations.
5. For Cohort B only: previous treatment with liposomal irinotecan for advanced or metastatic pancreatic cancer.
6. History of organ transplant requiring immunosuppression.
7. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
8. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count (ANC) < 1000 cells/mm3.
   2. Platelet count < 100,000 cells/mm3.
   3. Hemoglobin < 9 g/dL.
   4. Total bilirubin greater than two times the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   5. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. Alkaline phosphatase (ALP) levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   8. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
   9. Albumin <3.0.
   10. Ascites requiring paracentesis.

   Each site should use its own institution's ULN to determine eligibility.
9. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
10. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
11. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
12. Known hypersensitivity to any component of the study medication(s).
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to dosing for this study, except for testosterone-lowering therapy in men with prostate cancer or FDA-authorized drugs for the prevention and treatment of COVID-19.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women. A negative serum pregnancy test during screening and a negative pregnancy test within 72 hours prior to the first dose must be documented before study drug is administered to a female subject of child-bearing potential.
19. Any other cancer within the past 5 years that is progressing or requires active treatment, or any previous cancer treatment within the last 5 years that included gemcitabine or nab-paclitaxel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 8 weeks
  Response Criteria in Solid Tumors (RECIST) V1.1

SECONDARY OUTCOMES:
Objective response rate (ORR), Complete response (CR) rate, and Disease Control Rate (DCR) | 2 years
  Response Criteria in Solid Tumors (RECIST) V1.1
Overall Survival (OS) | 2 years
Quality of Life (QoL) | 2 years
  Patient Reported Outcomes (PROs) using the Functional Assessment of Cancer Therapy - Hepatobiliary Cancer (FACT-Hep) Questionnaire

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Chan Soon-Shiong Institute for Medicine, El Segundo, California
  - Hoag memorial Presbyterian Hospital, Newport Beach, California
  - Astera Cancer Care, East Brunswick, New Jersey
  - Avera Cancer Institute, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No